CLINICAL TRIAL: NCT05953376
Title: Empiric Calcium Versus Lab Based Treatment in Massive Transfusion Trauma Patients: A Feasibility Randomized Controlled Trial
Brief Title: Empiric Calcium in Massive Transfusion
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University of California, Irvine (Other)
Responsible Party: Principal Investigator, Jeffrey Nahmias, MD, Associate Professor of Surgery, University of California, Irvine
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 3115
Record Dates: First submitted 2023-07-11; First posted 2023-07-20 (Actual); Last update posted 2024-04-08 (Actual); Status verified 2024-04

CONDITIONS: Hemorrhage; Trauma; Hypocalcemia; Shock, Hemorrhagic
MeSH Terms: conditions — Hemorrhage; Wounds and Injuries; Hypocalcemia; Shock, Hemorrhagic | interventions — Calcium Gluconate; Calcium

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Empiric calcium administration (Experimental): Patients in this arm will receive 2g IV calcium with the initial transfusion
  Interventions: Drug: Calcium Gluconate
- No empiric calcium administration (No Intervention): Patients in this arm will only receive calcium supplementation based on routine ionized calcium levels and/or physician discretion

INTERVENTIONS:
Drug: Calcium Gluconate — There will be 2 study arms, one will receive 2g IV calcium with the initial transfusion and the other will only receive calcium supplementation based on routine ionized calcium levels and/or physician discretion.
  Other Names: Calcium
  Arms: Empiric calcium administration

SUMMARY:
Calcium helps blood to clot and thereby stop bleeding. Trauma patients who experience large volume blood loss often require blood transfusions and bleeding is the most common cause of death. The purpose of this study is to see if giving intravenous calcium immediately to patients who require large volume blood transfusion will decrease transfusion requirements, vasopressor use and mortality in bleeding trauma patients.

DETAILED DESCRIPTION:
Advancements in the area of transfusion and blood product administration have occurred with the use of viscoelastic assays and whole blood. However, as we resuscitate trauma patients with blood products, hypocalcemia is an inadvertent side-effect. Citrate within stored blood binds calcium, causing patients to have hypocalcemia. In addition, outside of transfusion related hypocalcemia there is an independent trauma/inflammation related mechanism for hypocalcemia in the trauma patient. Furthermore, Calcium is a critical component of the coagulation cascade, and therefore a highly important component of hemostatic resuscitation. Hall et al found that patients receiving 13 or more units of PRBCs had a much higher prevalence of severe hypocalcemia and at least one ionized calcium <1.0mmol/L. Kronstedt el al reported an association between hypocalcemia and mortality in trauma patients receiving massive transfusion. Despite evidence that hypocalcemia occurs with transfusion, and evidence that hypocalcemia in patients with hemorrhagic shock may be associated with increased mortality, there are no randomized controlled trials evaluating the administration of calcium in trauma resuscitation. Currently, the Joint Trauma System revised guidelines for damage control resuscitation from 2019 recommend administering 1g of calcium after the first unit of blood transfusion, and an additional 1g after no more than 4 units of blood administration. However, these recommendations are based on small cohort studies or retrospective studies. The purpose of this study is to evaluate the efficacy of early empiric intravenous calcium administration on transfusion requirements, vasopressor use and mortality in hemorrhaging trauma patients with initiation of a massive transfusion.

All trauma patients in which massive transfusion is initiated within 6 hours of arrival will be enrolled. Two study arms will be created, one will receive 2g IV calcium with the initial transfusion and the other will only receive calcium supplementation based on routine ionized calcium levels and/or physician discretion. All critical trauma activations will get a baseline ionized calcium as part of their initial labs.

ELIGIBILITY:
Inclusion Criteria:

* Trauma patients receiving massive transfusion protocol

Exclusion Criteria:

* Pregnancy
* Prisoners
* Known history of hypercalcemia
* Active hyperparathyroidism
* Hemophilia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-01 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Transfusion requirements | During first 24 hours of resuscitation
  Number of packed red blood cells, whole blood, fresh frozen plasma, platelets and cryo units given

SECONDARY OUTCOMES:
Mortality | 30-day mortality
  30-day mortality or until discharge (whichever is longer)
Vasopressor use | During first 24 hours of resuscitation
  Amount of vasopressor used within the first 24 hours measured in levophed equivalents

CONTACTS AND LOCATIONS:
Overall Officials: Jeffry Nahmias, MD, Principal Investigator — University of California, Irvine

REFERENCES:
- [Background] Hall C, Nagengast AK, Knapp C, Behrens B, Dewey EN, Goodman A, Bommiasamy A, Schreiber M. Massive transfusions and severe hypocalcemia: An opportunity for monitoring and supplementation guidelines. Transfusion. 2021 Jul;61 Suppl 1:S188-S194. doi: 10.1111/trf.16496. PMID 34269436
- [Background] Giancarelli A, Birrer KL, Alban RF, Hobbs BP, Liu-DeRyke X. Hypocalcemia in trauma patients receiving massive transfusion. J Surg Res. 2016 May 1;202(1):182-7. doi: 10.1016/j.jss.2015.12.036. Epub 2015 Dec 30. PMID 27083965
- [Background] Kronstedt S, Roberts N, Ditzel R, Elder J, Steen A, Thompson K, Anderson J, Siegler J. Hypocalcemia as a predictor of mortality and transfusion. A scoping review of hypocalcemia in trauma and hemostatic resuscitation. Transfusion. 2022 Aug;62 Suppl 1(Suppl 1):S158-S166. doi: 10.1111/trf.16965. Epub 2022 Jun 24. PMID 35748676
- [Background] Vettorello M, Altomare M, Spota A, Cioffi SPB, Rossmann M, Mingoli A, Chiara O, Cimbanassi S. Early Hypocalcemia in Severe Trauma: An Independent Risk Factor for Coagulopathy and Massive Transfusion. J Pers Med. 2022 Dec 28;13(1):63. doi: 10.3390/jpm13010063. PMID 36675724